CLINICAL TRIAL: NCT02255747
Title: Anal Dilatation for Infants and Children With Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jiexiong Feng, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anal Dilatation
Record Dates: First submitted 2014-09-28; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Constipation
Keywords: infants and children with constipation
MeSH Terms: conditions — Constipation | interventions — Lactulose

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- anal dilatation (Active Comparator)
  Interventions: Drug: Lactulose
- Oral Lactulose (Active Comparator)
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Lactulose

SUMMARY:
This study is to evaluate the effect of anal dilation in infants and children with constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and Children With Constipation
2. Postoperative infants and children with Hirschsprung's disease
3. Good compliance

Exclusion Criteria:

1. Infants and Children With Constipation
2. Poor compliance

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Daily stool times | two years

SECONDARY OUTCOMES:
The frequency of intestinal peristalsis waves | two years
The amplitude of intestinal peristalsis waves | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jiexiong, Feng, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China